CLINICAL TRIAL: NCT01911936
Title: A Phase I Study of LJM716 in Japanese Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLJM716X1101
Record Dates: First submitted 2013-07-24; First posted 2013-07-30 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2015-05

CONDITIONS: Neoplasms
Keywords: CLJM716,; Japanese patients,; Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LJM716 (Experimental)
  Interventions: Drug: LM716

INTERVENTIONS:
Drug: LM716

SUMMARY:
This study will evaluate safety and tolerability to estimate the MTDand/or recommended dose.

DETAILED DESCRIPTION:
This is a phase I, open-label, dose-escalation study to establish the MTD and/or RDE of LJM716 as single agent in Japanese patients that have advanced solid tumors. The study consists of a dose escalation part and a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the following indications:

   i) (Dose escalation part only): HER2 overexpressing locally advanced/ metastatic breast cancer or gastric cancer for which no effective treatment option exists:
   * For breast cancer: documented 3+ by immunohistochemistry, or amplification by in situ hybridization
   * For gastric cancer (including GE junction tumors): documented 3+ by immunohistochemistry, or 2+ by immunohistochemistry and amplification by in situ hybridization OR, ii) (Dose escalation part only): Recurrent or metastatic SCCHN regardless of HER2 status for which no effective treatment option exists OR, iii) Recurrent or metastatic ESCC regardless of HER2 status for which no effective treatment option exists
2. ECOG Performance Status of 0-2
3. Must have recovered from the adverse effects of any prior surgery, radiotherapy or other antineoplastic therapy. Alopecia and CTCAE Grade 1 peripheral neuropathy is acceptable.
4. Willingness and ability to comply with all study procedures
5. Written informed consent obtained prior to any screening procedures
6. During dose expansion part of the study, patients must have at least one measurable lesion as defined by RECIST v1.1 criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) in the dose escalation part | First cycle (28 days)

SECONDARY OUTCOMES:
Frequency and severity of adverse events, number of and reasons for | from informed consent till 30 days after end of treatment
LJM716 serum concentration-time- profile and estimated PK | up to 10 cycle (1 cycle = 28 days)
Tumor response according to RECIST 1.1 | every 2 months until end of treatment up to 2 years
Incidence of antibodies against LJM716 | up to 10 cycle ( 1cycle = 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Fukuoka

REFERENCES:
- [Derived] Takahashi S, Kobayashi T, Tomomatsu J, Ito Y, Oda H, Kajitani T, Kakizume T, Tajima T, Takeuchi H, Maacke H, Esaki T. LJM716 in Japanese patients with head and neck squamous cell carcinoma or HER2-overexpressing breast or gastric cancer. Cancer Chemother Pharmacol. 2017 Jan;79(1):131-138. doi: 10.1007/s00280-016-3214-4. Epub 2016 Dec 9. PMID 27942917
- See also: Results for CLJM716X1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14468